CLINICAL TRIAL: NCT00475527
Title: Helicobacter Pylori and Iron Deficiency: Prevalence of Association and Effect of Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: problem of accrual
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-HMO-CTIL
Record Dates: First submitted 2007-05-15; First posted 2007-05-21 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2009-01

CONDITIONS: Anemia, Iron-Deficiency; Helicobacter Pylori
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Omeprazole; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron only (No Intervention): Only iron therapy
- iron + HP therapy (Experimental): Iron + 'omeprazole,clarithromycin,amoxicillin (or metronidazole)
  Interventions: Drug: omeprazole,clarithromycin,amoxicillin (or metronidazole)

INTERVENTIONS:
Drug: omeprazole,clarithromycin,amoxicillin (or metronidazole)
  Arms: iron + HP therapy

SUMMARY:
Iron deficiency anemia (IDA) is a major health problem in children, effecting up to 20% of young children. Helicobacter pylori (HP) infection is also reported to be prevalent in children. Several large epidemiologic studies support an association between HP infection and lower iron stores. Other small studies suggest improvement in anemia following HP treatment.

We assume that the prevalence of HP infection in Israeli children diagnosed with IDA is high and that that adding therapy for HP in those children will improve the response to iron deficiency.

DETAILED DESCRIPTION:
This is a prospective randomized control study which will be conducted at six large ambulatory pediatrics clinics from the Jerusalem district. All of the children diagnosed with IDA would be eligible to join the study after informed consent will be obtained. Ethics committee approval is obtained. Analysis of stool samples will be carried out by the HP Stool antigen EIA (HpSA, Premier Platinum HpSA, Meridian Diagnostics inc, Cincinnati, OH, USA). All children enrolled will be treated with standard Fe therapy. Children with positive HpSA will be randomized, controlled for age and clinic, to receive or not receive antibiotics treatment. Assessment of response to iron therapy will be done at eight weeks later. The prevalence of HP infection in children with diagnosed with IDA would be reported. Statistical analysis will compare the baseline data between HP-positive and -negative children and the response to Fe between the three study groups.

ELIGIBILITY:
Inclusion Criteria:

* All of the children diagnosed with IDA at six large ambulatory pediatrics clinics from the Jerusalem district.
* The diagnosis of IDA would be defined as a low hemoglobin level in the presence of iron deficiency (low iron levels, high transferrin saturation and/or low ferritin).

Exclusion Criteria:

* Children with clinical symptoms fo Helicobacter Pylori, i.e. abdominal pain, peptic ulcer etc.
* Children with underlying chronic disease needing medical treatment.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To compare the raise in hemoglobin level between baseline and eight weeks later in Fe-supplemented and HP-positive children treated for HP infection and Fe-supplemented HP-positive children not treated for HP. | two years

SECONDARY OUTCOMES:
1. To determine the prevalence of HP infection in children with IDA in Israel, 2. To compare the demographic, clinical and laboratory findings between children diagnosed with IDA with/without HP infection. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Revel-Vilk, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel